CLINICAL TRIAL: NCT05187858
Title: A Phase I Open-Label Study of LNP3794 (BI3011441) in Subjects With NRAS/KRAS Mutated Advanced or Metastatic Refractory Solid Tumors
Brief Title: A Study of LNP3794 in Subjects With NRAS/KRAS Mutated Advanced or Metastatic Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LRP/LNP3794/2020/001
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: NRAS/KRAS Mutated Advanced or Metastatic Refractory Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LNP3794 (Experimental): Participants will receive LNP3794 orally once daily at different doses in 28 day cycles on a continuous basis
  Interventions: Drug: LNP3794

INTERVENTIONS:
Drug: LNP3794 — LNP3794 capsules administered orally once daily

SUMMARY:
This is a Phase I, open-label, dose escalation study of LNP3794 (BI3011441) in subjects with NRAS/KRAS mutated advanced or metastatic refractory solid tumors. The purpose of this study is to evaluate the safety/tolerability, pharmacokinetic and pharmacodynamic profile of the orally administered LNP3794 (BI3011441) as monotherapy at selected dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years of age
2. Pathologically documented, locally-advanced or metastatic solid malignancy with NRAS or KRAS mutation
3. At least one target lesion that can be measured per RECIST version 1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Adequate organ function (bone marrow, hepatic, renal, cardiovascular)
6. Documented disease progression despite appropriate prior standard therapies or subjects for whom no standard therapy exists for their tumor type and disease stage
7. Reproductive criteria (as defined in the protocol)

Exclusion Criteria:

1. Subjects with symptomatic central nervous system (CNS) metastases
2. History of another primary malignancy, with the exception of locally excised nonmelanoma skin cancer and carcinoma in situ of uterine cervix
3. Known active hepatitis B infection or hepatitis C infection
4. Known pre-existing interstitial lung disease
5. Known diagnosis of human immunodeficiency virus (HIV) infection
6. History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy; or known risk factors for RVO or central serous retinopathy
7. Any severe and/or uncontrolled medical conditions or other conditions that, in the opinion of the Investigator, Sponsor, or contract research organization, could affect the subject's participation in the study
8. Impaired cardiac function or clinically significant cardiac diseases
9. Previous treatment with RAS or MEK targeting agents
10. Chemotherapy, biologic therapy, immunotherapy, radiotherapy, or investigational agents within 5 half-lives or within 4 weeks (whichever is longer) prior to administration of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities (DLTs) at each dose level during the first cycle | up to Day 28
  Dose limiting toxicities will be evaluated through the first cycle (each cycle is 28 days)

SECONDARY OUTCOMES:
Number of subjects with DLTs during the entire on-treatment period | up to 2 years
  Dose limiting toxicities will be evaluated through the entire on-treatment period
Number of subjects with Grade ≥3 treatment-related adverse events (AEs) | up to 2 years
  Grade ≥3 treatment-related adverse events will be evaluated through the entire on-treatment period
Number of subjects with treatment-related AEs at each dose level | up to 2 years
  Treatment-related AEs at each dose level will be evaluated through the entire on-treatment period
Maximum Plasma Concentration (Cmax) of LNP3794 | Cycle 1 (each cycle is 28 days) Day 1 and Day 14
  Cmax is the maximum observed plasma concentration.
Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) | Cycle 1 (each cycle is 28 days) Day 1 and Day 14
  AUC[0-last] is the measure of plasma drug concentration from time zero to the time of last quantifiable concentration.
Area under the concentration-time curve from time zero to the end of dosing interval (AUC[0-tau]) | Cycle 1 (each cycle is 28 days) Day 1 to 2 and Day 14 to 15
  AUC[0-tau] is the measure of plasma drug concentration from time zero to the end of dosing interval.
Time to maximum concentration (Tmax) | Cycle 1 (each cycle is 28 days) Day 1 and Day 14
  Tmax is the time to reach maximum plasma concentration.

OTHER OUTCOMES:
Change from baseline in pERK levels | Baseline and Cycle 1 (each cycle is 28 days) Day 14
  Change from baseline in pERK levels will be evaluated
Objective response rate (ORR) and disease control rate (DCR) | up to 2 years
  Objective response rate (ORR) and disease control rate (DCR) will be determined using response evaluation criteria in solid tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanajay Bakhle, MD, Study Chair — Lupin Limited
Locations (4):
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- Amsterdam UMC, Amsterdam, Netherlands
- United Kingdom (2):
  - Sarah Cannon Research Institute, London
  - The Christie NHS Foundation, Manchester